CLINICAL TRIAL: NCT04491253
Title: Efficacy of a Social Support Intervention in Adults for Self-management of Type 2 Diabetes Mellitus
Brief Title: Social Support Intervention for Self-management of Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-04
Record Dates: First submitted 2020-07-24; First posted 2020-07-29 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Nursing Outcomes Classification Terminology; Self-management; Social support
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention is defined as informational support (transmission of information for health care, knowledge of DM2, nutrition, physical activity), instrumental (physical care) and emotional (management of anxiety, empowerment and decision-making).
  Interventions: Behavioral: Social support for diabetes self-management
- Control (No Intervention): Control group will receive usual care treatment at the diabetes mellitus nursing consultation in primary care.

INTERVENTIONS:
Behavioral: Social support for diabetes self-management — Four individualized intervention sessions, every two weeks with a duration of 40 minutes.
  Arms: Intervention

SUMMARY:
This study will assess the effect of a social support intervention for self-management of type 2 diabetes mellitus (DM2) in adults. This intervention is based on a medium-range nursing theory of individual and family self-management. Findings will be evaluated using the nursing outcomes "self-management: diabetes" and "social support" from the Nursing Outcomes Classification (NOC).

DETAILED DESCRIPTION:
Diabetes mellitus is responsible for 1.6 million deaths a year, becoming one of the world's 21st century health emergencies.

DM2 is the most frequent form of diabetes, accounting for 90% of all cases of this chronic condition. If this trend continues, by 2045 about 693 million people will have diabetes.

People with chronic diseases have changing perspectives, in addition to suffering physical alterations, their psychological, emotional and social state is also compromised, presenting themselves as a need to modify lifestyle to improve prognosis, facing alterations in the ability to socialize and with death or a great loss. Few studies comprehensively address these dimensions.

The literature reports that DM2 self-control has a direct effect in improving clinical results, reducing complications and quality of life. Therefore, the patient must make multiple decisions every day regarding diet, physical activity, glucose control, and medication compliance.

However, intervention studies that seek to improve self-management behaviors in people with DM2 are characterized by emphasizing the transmission of knowledge and establishing compliance with prescribed treatments, but they do not address social and emotional elements such as social support. Additionally, most of these interventions do not show the use of theoretical models that provide explanations of human responses to disease and other phenomena important to practice.

Studies using the Nursing Outcomes Classification to assess the effect of social support interventions are scarce.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years with a diagnosis of DM2, attending the outpatient diabetes consultation at the health care institution.
* Initial score less than or equal to 3 on the NOC outcomes: self-management: diabetes and social support.

Exclusion Criteria:

* People with a score <30 on the cognitive mini mental test.
* Other comorbidities reported by the patient or in the medical history that limit receiving the intervention (example: hearing loss, deafness, Alzheimer's disease).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Self-management: diabetes | 2 months
  NOC outcome. Personal actions to manage diabetes, its treatment, and to prevent complications. Indicators of participation in self-management behaviors, specifically healthy eating, physical exercise, glucose monitoring and symptom management. This outcome will be evaluated by a Likert scale, being 1 the worst score and 5 best score.

SECONDARY OUTCOMES:
Social support | 2 months
  NOC outcome. Reliable assistance from others. Indicators of emotions, stress, communication, decision-making, empowerment, trust, support groups and networks. This outcome will be evaluated by a Likert scale, being 1 the worst score and 5 best score.

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Canon Montanez, PhD, Study Director — Universidad de Antioquia
Locations (1):
- Universidad de Antioquia, Medellín, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garizábalo-Dávila CM, Rodríguez-Acelas AL, Cañon-Montañez W. Soporte social enfocado a personas con diabetes: una necesidad desde enfermería. Rev Cuid. 2019; 10(1): e697. http://dx.doi.org/10.15649/cuidarte.v10i1.697
- [Background] Garizábalo-Dávila CM, Rodríguez-Acelas AL, Mattiello R, Cañon-Montañez W. Social Support Intervention for Self-Management of Type 2 Diabetes Mellitus: Study Protocol for a Randomized Controlled Trial. Open Access Journal of Clinical Trials. 2021;13:37-43 https://doi.org/10.2147/OAJCT.S314030